CLINICAL TRIAL: NCT02824341
Title: Exploration of the Reward System by Functional MRI in Parkinson's Disease Patients With and Without REM Sleep Behavior Disorder
Acronym: MP-TCSP-IRMf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Neurodis Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0270; 2015-A00761-48 (Other: 2015-A00761-48)
Record Dates: First submitted 2016-06-24; First posted 2016-07-06 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Parkinson's Disease; REM Sleep Behavior Disorder
Keywords: Parkinson 's disease; REM sleep behavior disorder; Reward system; Functional MRI
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder | interventions — Magnetic Resonance Imaging

ARMS (3):
- Parkinson's disease patients with RBD (Other): The investigators hypothesize that PD patients with RBD have a more severe dysfunction of the reward system (hypoactivation of the meso-cortico-limbic pathway) than patients without RBD, explaining their susceptibility to ICD when exposed to high doses of dopaminergic treatment.
  Interventions: Device: fMRI
- Parkinson's disease without RBD (Other): The investigators hypothesize that PD patients with RBD have a more severe dysfunction of the reward system (hypoactivation of the meso-cortico-limbic pathway) than patients without RBD, explaining their susceptibility to ICD when exposed to high doses of dopaminergic treatment.
  Interventions: Device: fMRI
- Healthy volunteers (Other): The investigators hypothesize that PD patients with RBD have a more severe dysfunction of the reward system (hypoactivation of the meso-cortico-limbic pathway) than patients without RBD, explaining their susceptibility to ICD when exposed to high doses of dopaminergic treatment.
  Interventions: Device: fMRI

INTERVENTIONS:
Device: fMRI

SUMMARY:
Up to 60% of Parkinson's Disease (PD) patients suffer from REM sleep behavior disorder (RBD), a parasomnia. This disorder is thought to be related to a dysfunction of limbic system and brainstem.

Impulse control disorders (ICD) are found in about 14% of PD patients taking dopaminergic drugs. These disorders are thought to be related to a dysfunction of meso-cortico-limbic pathways which belong to the so-called "reward system".

A strong link was found between these two disorders and therefore the investigators believe that RBD is associated with impaired reward system.

The main objective of this study is to evaluate differences in brain activation between PD patients with and without RBD.

The investigators hypothesize that PD patients with RBD have a more severe dysfunction of the reward system (hypoactivation of the meso-cortico-limbic pathway) than patients without RBD, explaining their susceptibility to ICD when exposed to high doses of dopaminergic treatment.

DETAILED DESCRIPTION:
Type of study: Prospective, case control study.

Number of centers: 2 (Clermont-Ferrand and Vichy)

Patients :

The study will be performed in 75 subjects (25 PD patients with RBD, 25 PD patients without RBD and 25 healthy volunteers, age-and sex-matched without any contraindications to perform an MRI)

Study Performance :

During the first visit (J0, inclusion visit, 3 hours), each subject will perform a clinical and neurological examination (MDS-Unified Parkinson Disease Rating scale (MDS-UPDRS)) and neuropsychological assessment (depression by the Beck Depression Inventory (BDI); apathy by the Lille Apathy Rating Scale (LARS), impulsivity by the Urgency, lack of Premeditation, lack of Perseverance, Sensation Seeking scale (UPPS)) Eligible patients will be welcomed in a subsequent visit at the MRI department for the functional MRI (J0+1week, 1 hour). This session will be of about 45 minutes. The reward system was explored using an experimental task during functional Magnetic Resonance Imaging (fMRI). The name of this task is the"monetary incentive delay task".

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease (UK Parkinson's Disease Society Brain Bank Criteria)
* men or women 45 to 80 years old
* diagnosis of RBD made with polysomnographic recording

Exclusion Criteria:

* Previous history of psychosis or psychiatric disease
* History of stroke or vascular lesion on MRI.
* pregnant women

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
BOLD signal variation in each region of interest | at week 1
  BOLD signal variation in each region of interest (ventral tegmental area, accumbens nucleus, limbic cortex, prefrontal cortex) at the time of realisation of fMRI.

SECONDARY OUTCOMES:
Reaction time to the task | at week 1
Performance score to the task | at week 1
Hoehn et Yahr score | at week 1
The Unified Parkinson Disease Rating scale (MDS-UPDRS) score | at week 1
The Beck Depression Inventory score | at week 1
The Lille Apathy Rating Scale score | at week 1
The impulsivity score by the Urgency | at week 1

CONTACTS AND LOCATIONS:
Overall Officials: Franck DURIF, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France